CLINICAL TRIAL: NCT00186966
Title: A Randomized Phase III Study of the Treatment of Children and Adolescents With Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: Treatment of Children and Adolescents With Refractory or Relapsed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dutch Childhood Oncology Group (Other)
Collaborators: International BFM Study Group (Network); St. Jude Children's Research Hospital (Other)
Responsible Party: Prof. G.J.L. Kaspers, MD PhD / Principal Investigator, Dutch Childhood Oncology Group, the Hague, the Netherlands
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIAL; TRIAL Relapsed AML 2001/01
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; Cytarabine; Daunorubicin; Etoposide; Thioguanine; Cyclophosphamide; Busulfan; Melphalan; Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FLAG (Other)
  Interventions: Drug: Fludarabine, Cytarabine, Liposomal daunorubicin (DaunoXome); Drug: Etoposide, Thioguanine, Cyclophosphamide, Busulfan, Melphalan; Procedure: Hematopoietic stem cell transplant; Radiation: Total body irradiation
- FLAG and LP Dox (Other)
  Interventions: Drug: Fludarabine, Cytarabine, Liposomal daunorubicin (DaunoXome); Drug: Etoposide, Thioguanine, Cyclophosphamide, Busulfan, Melphalan; Procedure: Hematopoietic stem cell transplant; Radiation: Total body irradiation

INTERVENTIONS:
Drug: Fludarabine, Cytarabine, Liposomal daunorubicin (DaunoXome) — See Detailed Description section for details of treatment interventions.
Drug: Etoposide, Thioguanine, Cyclophosphamide, Busulfan, Melphalan — See Detailed Description section for details of treatment interventions.
Procedure: Hematopoietic stem cell transplant — See Detailed Description section for details of treatment interventions.
Radiation: Total body irradiation — See Detailed Description section for details of treatment interventions.

SUMMARY:
This is an international multicenter open label randomized phase III trial in children with relapsed and refractory acute myeloid leukemia (AML) such a disease. The main purpose of this study is to determine the efficacy and toxicity of liposomal daunorubicin when added to fludarabine, ara-C and G-CSF(FLAG) in children with relapsed and refractory AML.

DETAILED DESCRIPTION:
Secondary objectives of this trial are:

* To determine the toxicity of liposomal daunorubicin when added to FLAG, in terms of mucosal toxicity, bone marrow aplasia, short- and long-term cardiotoxicity and other side effects as compared to patients treated with FLAG only.
* To determine the long-term clinical outcome prospectively in a large group of children with refractory and relapsed acute myeloid leukemia.
* To determine the changes in minimal residual disease over time, and the prognostic significance of minimal residual disease determined at various time-points.
* To determine the relation between in vitro cellular drug resistance and clinical and cell biological features, minimal residual disease and clinical outcome in this patient group
* To determine the pharmacokinetics of liposomal daunorubicin in relation to its toxicity and efficacy

Reinduction treatment will be done with 2 courses of combination chemotherapy, with FLAG (fludarabine, ara-C and G-CSF) in both courses as standard treatment. In the first course there will be a randomisation for liposomal daunorubicin (DaunoXome®) to be added or not. The second course should always concern FLAG. If patients have > 20% of blasts in the bone marrow after the 1st course, or if they are not in complete remission (CR) after the 2nd course, they will go off protocol. Patients in CR after reinduction treatment can immediately proceed to stem cell transplantation. Consolidation chemotherapy should be given if SCT is delayed. A 3rd course of intensive chemotherapy (VP16 and continuous infusion with cytarabine) is the general recommendation. In selected patients, a low intensity consolidation may be preferred, and such a schedule is described as well. The type of SCT is based on the risk-group. Preferably, a matched sibling donor (MSD) SCT is performed. If a MSD is not available all patients are candidates for a matched unrelated donor (MUD) SCT. If a MUD is also not available, patients with primary refractory disease, early relapse (within 1 year from diagnosis), or greater than or equal to 2nd relapse, are candidates for the more experimental haplo-identical donor (HID) SCT in view of the dismal prognosis. However, patients with a late relapse (>1 year from initial diagnosis) have a better prognosis and should be offered an autologous SCT if a MSD or MUD SCT is not possible. Only in case of autologous SCT, maintenance treatment and/or adjuvant immunotherapy could be considered.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents less than eighteen years of age at start of chemotherapy.
* Subject has one of the following: Primary refractory AML, first relapsed AML, second or subsequent relapsed AML and was not previously treated according to this particular protocol
* Subjects with a combined relapse, or an isolated extramedullary relapse, or a bone marrow relapse are eligible, also for randomization.

Exclusion Criteria:

* Symptomatic cardiac dysfunction.
* Inadequate performance score.
* Any other organ dysfunction that will interfere with the administration of the therapy.
* FAB type M3

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 394 (Actual)
Dates: Start 2002-03; Primary Completion 2009-04 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Response Rate | 8-9 years

SECONDARY OUTCOMES:
Toxicity between two arms | 8-9 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Rubnitz, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Result] Kaspers J, Zimmermann M, Fleischhack G, Tamminga R, Gibson B, Armendariz H, Dworzak M, Ha S, Hovi L, Maschan A, Philippe N, Razzouk B, Rizzari C, Smisek P, Smith O, Stark B, Will A, Creutzig U. Relapsed Acute Myeloid Leukemia in Children and Adolescents: Interim Report of the International Randomised Phase III Study Relapsed AML 2001/01. 2006 ASH Annual Meeting Abstracts 108: 2013.
- See also: St. Jude Children's Research Hospital — http://www.stjude.org